CLINICAL TRIAL: NCT05543473
Title: Effect of Vestibular Rehabilitation Therapy on Patients With Brain Radiological Findings That Affect Balance Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Nasser Fahmy, Resident doctor at audio-vestibular medicine unit sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-13
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Brain Vascular Insult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients with brain radiological findings that affect balance functions
  Interventions: Other: Vestibular Rehabilitation Therapy

INTERVENTIONS:
Other: Vestibular Rehabilitation Therapy — an exercise-based treatment program designed to promote vestibular adaptation and substitution. The goals of VRT are to enhance gaze stability, to enhance postural stability, to improve vertigo, and to improve activities of daily living. VRT facilitates vestibular recovery mechanisms: vestibular adaptation, substitution by the other eye-movement systems, substitution by vision, somatosensory cues, other postural strategies, and habituation

SUMMARY:
Occurrence of cerebrovascular diseases, particularly of cerebral small vessel disease (SVD), appears to play some role in the development of gait and balance impairment . Beside small vessel disease , stroke is one of the most common cause of long-term adult disability leading to cognitive and motor function impairments. Particularly, gait and balance disorders that may contribute to immobility and falls.

The design of personalized rehabilitation protocols, focused on the recovery of dynamic balance ability would be fundamental to reduce these deficits and consequently, the risk of falling, thus improving patients' quality of life. Vestibular rehabilitation therapy (VRT) is an exercise-based treatment program designed to promote vestibular adaptation and substitution. The goals of VRT are to enhance gaze stability, to enhance postural stability, to improve vertigo, and to improve activities of daily living. VRT facilitates vestibular recovery mechanisms: vestibular adaptation, substitution by the other eye-movement systems, substitution by vision, somatosensory cues, other postural strategies, and habituation .

ELIGIBILITY:
Inclusion Criteria:

* Age: from 40 years to 60 years old.
* Sex: males and females.
* Can withstand and willing to undergo repeated CDP trials.
* No evidence of orthopedic problems, neurological or cardiovascular diseases. - No history of any disease required to give treatment that could affect results.

Exclusion Criteria:

* Geriatric population , above age 60 years old.
* Patients with orthopedic problems , neurological or cardiovascular diseases.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of change in balance function | 3 months after the end of Vestibular rehabilitation therapy
  The computerized dynamic posturography sensory organization test (CDP-SOT)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmad H, Cerchiai N, Mancuso M, Casani AP, Bronstein AM. Are white matter abnormalities associated with "unexplained dizziness"? J Neurol Sci. 2015 Nov 15;358(1-2):428-31. doi: 10.1016/j.jns.2015.09.006. Epub 2015 Sep 4. PMID 26412160
- [Background] Alcock L, O'Brien TD, Vanicek N. Association between somatosensory, visual and vestibular contributions to postural control, reactive balance capacity and healthy ageing in older women. Health Care Women Int. 2018 Dec;39(12):1366-1380. doi: 10.1080/07399332.2018.1499106. Epub 2018 Nov 5. PMID 30395787
- [Background] Alyono JC. Vertigo and Dizziness: Understanding and Managing Fall Risk. Otolaryngol Clin North Am. 2018 Aug;51(4):725-740. doi: 10.1016/j.otc.2018.03.003. Epub 2018 May 24. PMID 29803531
- [Background] Ekvall Hansson E, Pessah-Rasmussen H, Bring A, Vahlberg B, Persson L. Vestibular rehabilitation for persons with stroke and concomitant dizziness-a pilot study. Pilot Feasibility Stud. 2020 Sep 30;6:146. doi: 10.1186/s40814-020-00690-2. eCollection 2020. PMID 33005434